

## **FRAILCLINIC**

## Study Title:

# FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFERRENT CLINICAL SETTINGS INTERVENTIONAL PHASE

Protocol identifying number: 20131208

## **Confidentiality Statement:**

This document contains confidential information that must not be disclosed to anyone other than the Sponsor, the Investigator Team, Regulatory Authorities, and members of the Ethics Committee.

Sponsor: FUNDACIÓN PARA INVESTIGACION BIOMÉDICA DEL HOSPITAL UNIVERSITARIO DE GETAFE

Project Leader: Prof. Leocadio Rodríguez Mañas

Medical monitor: Prof. Leocadio Rodríguez Mañas.

Email: leocadio.rodriguez@salud.madrid.org

Fax: 0034 916247305

Study promoted by DG SANCO "HEALTH-2013



## **TABLE OF CONTENTS**

| <u>1</u> | <u>AI</u> | BREVIATIONS | <u> 5</u> |
|---|---|---|---|
| <u>2</u> | <u>IN</u> | TRODUCTION | 6 |
| | 2.1 | BACKGROUND INFORMATION: | |
| | 2.2 | RATIONALE OR JUSTIFICATION | . 7 |
| <u>3</u> | OI | BJECTIVES | 9 |
| _ | 3.1 | PRIMARY OBJECTIVE: | |
| | 3.2 | SECONDARY OBJECTIVES: | . 9 |
| <u>4</u> | ΩI | UTCOMES | 11 |
| <b>I</b> | 4.1 | PRIMARY OUTCOMES: | |
| | 4.2 | SECONDARY OUTCOMES: | |
| _ | СТ | TUDY DESIGN | |
| <u>5</u> | | | |
| <u>6</u> | | LEGIBILITY | |
| | | NCLUSION CRITERIA: | |
| | 6.2 | EXCLUSION CRITERIA: | 15 |
| <u>7</u> | <u>RI</u> | ECRUITMENT | 16 |
| | 7.1 | INFORMED CONSENT AND ELEGIBILITY CRITERIA | |
| | 7.2 | RANDOMIZATION | 17 |
| | 7.3 | SAMPLE SIZE | 17 |
| | 7.4 | STATISTICAL ANALYSIS | 18 |
| <u>8</u> | <u>IN</u> | TERVENTION AND CONTROL | 20 |
| | 8.1 | CONTROL GROUP | 20 |
| | 8.2 | INTERVENTION GROUP | 20 |
| <u>9</u> | AS | SSESMENTS DURING THE STUDY | 21 |
| | 9.1 | BASELINE EVALUATION (visit 0= FIRST VISIT) | |
| | 9.2 | EVALUATION AT DISCHARGE FROM THE SPECIFIC CLINICAL SETTING | 22 |
| | 9.3 | EVALUATION AT 3 MONTHS OF DISCHARGE | 23 |
| | 9.4 | EVALUATION AT 12 MONTHS OF DISCHARGE | 23 |
| | 9.5 | END OF THE STUDY EVALUATION | 23 |
| 10 | 0. EC | ONOMIC EVALUATION | 26 |



| 11. APPENDIX | 30 |
|----------------|----|
| 12. REFERENCES | |



## **SIGNATURE PAGE**

## STUDY TITLE: FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE OLDER PATIENTS IN DIFFERENT CLINICAL SETTINGS

## **STUDY CODE:** FRAILCLINIC

| I confirm I have read and understand the prostudy according to what is recorded on it and | | |
|---|---|---|
| SPONSOR | | DATE |
| PROJECT COORDINATOR | | DATE |
| Prof. Leocadio Rodríguez Mañas | | |
| SCIENTIFIC COORDINATOR | DATE | |
| Name | | |
| Site | | |



## 1 ABREVIATIONS

| ADL | Activities of Daily Living |
|---------|--------------------------------------------------------|
| AE | Adverse event |
| GDS | GeriatricDepresionScale |
| FC | Fried's Criteria |
| EC | Ethics Committee |
| eCRF | Case Report Form |
| GCP | Good Clinical Practice |
| EQ-5D | EuroQolfive-dimensional (EQ-5D) |
| CRO | Contract Research Organization |
| IADL | Instrumental Activities of Daily Living |
| INE | Instituto Nacional de Estadística (Spain) |
| ICF | InformedConsentForm |
| MMSE | Minimental State Examination |
| SPPB | Short Physical Performance Battery |
| PASE | Physical Activity Scale for the Elderly |
| CAM | Confusion Assessment Method |
| ICER | Incremental cost-effectiveness ratio |
| PI | Principal Investigator |
| HUG-GRT | Hospital Universitario de Getafe-Servicio de Geriatría |



## 2 INTRODUCTION

## 2.1 BACKGROUND INFORMATION:

Disability is the main consequence of the concurrence of three conditions in old people: the ageing process, lifestyle processes and health-related conditions.

As it has been the case with other relevant organizations and bodies, in its 2012 Ageing report, the European Commission and the Economic Policy Committee stated that coping with the challenge posed by an ageing population and a trend toward increases in agerelated spending will require determined policy action in Europe, particularly in: (a) reforming pension, health care and long-term care systems, and (b) the reduction of disability and dependence through appropriate action with a special focus in fighting against disability (DG ECFIN & AWG, 2012).

Disability is usually preceded by a state characterized by a decreasing capacity to respond to demands, caused by diminishing functional reserve. This condition has been named frailty, a disorder that may precede by several years the development of disability (1) and other clinical outcomes. When the frailty threshold has been surpassed and disability has emerged, recovery from disability is unlikely (2), especially as the age of the patient, the degree of disability or its duration increase (3). In contrast, frailty is reversible, as it has been shown both spontaneously (4, 5) and by interventions based on physical exercise (6).

Moreover, and differently from chronic disease, the predictive capacity of frailty for adverse outcomes increases as the age of the population increases (8) becoming the most common condition leading to death among community-dwelling older persons, followed by organ failure (21.4%), cancer (19.3%) and dementia (13.8%) of dying.

The aim of the present study is to assess the feasibility and effectiveness of programs designed to detect and manage frail older patients in high risk clinical settings, and to avoid functional impairment and other associated adverse outcomes.



## 2.2 RATIONALE OR JUSTIFICATION

The prevalence of frailty in people older than 65 years is high, ranging from 7 to 16.3 %, and this increases with age (1, 9, 10).

The most accepted approach defines frailty as "an age-associated biological syndrome characterized by a decrease in biological reserve and resistance to stress, due to a decline in several physiological systems, placing the individual in a special risk category when facing minor stressors and associated with poor outcomes (disability, death and hospitalization)" (11-14).

Frailty is an established and credible concept which provides the framework for the relationships between ageing, disease, vulnerability, disability, and dependency (15). with its high prevalence in older people and its potential reversibility, make frailty the perfect target to overcome the challenge of disability in older adults (16).

The challenge for Health Systems is develop strategies to detect this syndrome and the prevention the functional decline and disability. As a consequence, a complementary strategy is needed, supporting clinicians to provide personalized, comprehensive continuity of care (17).

Older frail patients are prone to develop functional impairments, to be institutionalized and to die early. Additionally, they use Health and Social facilities much more frequently than their same-age counterparts, being at high risk for mis-, under- and over management. Some of these specific needs are covered by classical Geriatric facilities available in many European Hospitals. But these facilities only attend to 10-15% of all the frail older patients that are being seen and managed by other parts of the health care systems (14)

It has been largely recommended that programs must not only identify at-risk patients so that they may benefit from specialized management, but they must also target the process of care (Lafont E et al., JNHA 2011) to 1) provide the best-fitted models of care to their needs, and 2) adapt the management of their diseases and conditions (cancer, major surgery, heart disease, etc.) to their special features (18). In this regard, recent publications have stated that this approach should be standard practice, and is supported by a wealth of evidence (19), mainly in frail elderly patients being attended in some specific high risk settings as described in our proposal (20-23).



FRAILCLINIC project includes two consecutives phases: the first one focus on detection and quantification of frailty (observational phase) and the second phase focus on management of frail patients by an integrate model of geriatric care (interventional phase). In the observational phase we have evaluated the prevalence of frailty, the success of a program for detection frail patients in high risk clinical settings, tools commonly used for assessment of frailty and causes of no implementation. In the interventional phase we will analyse the effect of the performance of a geriatrician agreed with the treating physician/surgeon of the patient in these clinical settings comparing with the traditional performance.



## 3 OBJECTIVES

## 3.1 PRIMARY OBJECTIVE:

To assess the feasibility and effectiveness of programs designed to detect and manage frail older patients in high risk clinical settings, and to avoid functional impairment and other associated adverse outcomes. These high risk settings will be medical wards (cardiology, oncology or nephrology), major surgery wards and Emergency rooms.

## **3.2 SECONDARY OBJECTIVES:**

- Determine the feasibility of implementing clinical and therapeutic approach to geriatric physician in elderly patients in high risk clinical settings
- Determine disability by evaluating basic and instrumental activities of daily living in frail elderly patients treated in high risk clinical settings.
- o Establish functional status in frail elderly people seen in high risk clinical settings.
- Evaluate quality of life through an instrument validated in frail patients seen in high risk clinical settings.
- o Establish mortality ratio in frail patients included in high risk clinical settings.
- Obtain the rate of re-hospitalization in frail patients seen in high risk clinical settings.
- Determine the average stay of hospitalization in frail elderly patients treated in high risk clinical settings.
- Obtain the rate readmission to emergency room and hospitalization in frail older patients treated in high risk settings.
- Determine the average stay of hospitalization in frail elderly patients treated in high risk clinical settings.
- o Determine the rate of delirium in frail elderly patients in high risk settings.
- Obtain the rate of health-care associated infections in frail older patients seen in high risk settings.
- Determine the rate of polypharmacy in frail older patients seen in high risk settings.
- Establish the secondary institutionalization rate accordingly to decline the functional status in frail elderly patients in high risk settings.



- Determine the need for a caregiver as a result of decline the functional status in frail older people in high risk settings.
- o Establish the caregiver burden in hospitalized frail patients on high risk settings.
- Establish the secondary institutionalization rate accordingly to decline the functional status in frail elderly patients in high risk settings.
- Determine the need for a caregiver as a result of decline the functional status in frail older people in high risk settings.
- Establish caregiver burden of frail elderly patients seen in high risk settings.
- To evaluate the cost-effectiveness of the intervention compared with usual care from the perspective of society and the health system.
- o To evaluate the cost-utility of the intervention compared with usual care.



## 4 OUTCOMES

### 4.1 PRIMARY OUTCOMES:

- **1. Disability:** It was measured by the Barthel Index for basic Activities of Daily Living and the Lawton index for instrumental activities of daily living.
- 2. **Functional status and performance-based measures:** Functional status and performance-based measures: Is measured by Short Physical Performance Battery (SPPB), Physical Activity Scale for the Elderly (PASE SCALE).
- 3. **Quality of Life**: Quality of life was assessed by self-reported questionnaire EuroQL 5D 5L. It will be measured during admission to hospital and follow-up.
- 4. **Geriatrician Intervention**: The impact of their intervention is measured by quantifying in a register any additional tests requested and medical advice by other specialists.

## **4.2 SECONDARY OUTCOMES:**

**Prevalence of Delirium:** The delirium cases are detected by Confusion Assessment Method (CAM) scale.

**Cognitive Impairment:** Will be measured by the Mini Mental State Examination (MMSE) in the initial assessment.

**Depression**: will be assessed using the Geriatric Depression Scale in the baseline assessment.

**Health-care associated infections**: Acquired during hospitalization start.

**Geriatric Syndromes**: The geriatric evaluation including the following aspects: clinical, functional, mental and social.

Comorbidity: Will measured at initial assessment thorough Charlson index

**Nutritional Status**: Will measured at initial assessment thorough the Mini Nutritional Assessment and body Mass index.

**Polypharmacy**: Defined as five or more prescription drugs.

**Mortality rate**: Number of deaths during follow-up. It is calculated using official report of the National Statistics Institute (INE).

**Average stay hospitalization**: Average length of stay of stay all discharges. We will obtain from Hospital Admissions service.



**Hospitalization Rate in Emergency room**: Number of hospital admissions over the total of patients admitted in the hospital.

**Readmission rates**: Number of readmissions during of follow-up period. I will get the data in Hospital Admissions Service.

**Institutionalization:** Number of patients referred to nursing home after discharge or at any time during follow-up. This information is obtained directly from patients or their relatives.

**Requirement of caregiver**: Number of patients who require a caregiver after hospital discharge.

Caregiver burden: Will be used Zarit Scale for assessing caregiver burden

**Cost-effectiveness**: The incremental cost-effectiveness ratio (ICER) was assessed by measuring the difference in health outcomes per unit cost.

**Cost-utility**: is measured using the QALY (unit of measurement of preferences of individuals with regard to the quality of life that has occurred through a health intervention, combined with the years earned for a given health state).



## **5 STUDY DESIGN**

This trial is designed as a randomised, multicenter, phase III trial to evaluate the feasibility and viability of clinical and therapeutic approach frail older people in high risk clinical settings (Emergency room, General Surgery, Oncology, Cardiology, and Nephrology). Patients will be randomized on a 1:1 basis to receive either usual treatment or usual treatment plus geriatric interventions.

The patients will be recruitment in Spain, Italy and United Kingdom. In Spain will be included the following centres: Hospital Universitario de Getafe (Madrid), Hospital Universitario Central de Asturias Monte Naranco (Asturias); In Italy: Ospedale San Raffaele (Rome), Universitat'Cattolica del Sacro Cuore(Roma), in United Kingdom: (Cardiff University and other one to be determined)According to feasibility in each centre will be recruitment patients from differents clinical settings. See Table No 1



Table 1. Recruitment distribution of patients according to hospital and setting

| Hospital | Setting |
|------------------------------------------|-------------------|
| | Emergency room |
| Hospital Universitario de Getafe. | Cardiology ward |
| ladrid - Spain) | Elective Surgery |
| | Emergency Surgery |
| ospital Universitario Monte Naranco. | Oncology |
| (Asturias - Spain) | Elective Surgery |
| (Asturias - Spairi) | Emergency Surgery |
| Professor Sinclair | Emergency room |
| (England – United Kingdom) | Cardiology Ward |
| (England – Officed Kingdom) | Elective Surgery |
| | Emergency room |
| Cardiff University (Wales - Reino Unido) | Nephrology ward |
| | Elective Surgery |
| Ospedale San Raffaele | |
| (Rome - Italy) | Cardiology Ward |
| Universita' Cattolica del Sacro Cuore | Emergency Room |
| (Rome - Italy) | Cardiology Ward |
| | Elective Surgery |



## **6 ELEGIBILITY**

## **6.1 INCLUSION CRITERIA:**

Participants must meet all of the following inclusion criteria to be eligible to register for this trial: older than 75 years old diagnosed of frailty, according to Fried's Criteria, if is not possible to use the Fried Scale, FRAIL Scale will be used.

## **6.2 EXCLUSION CRITERIA:**

- Do not able to give informed consent.
- Participants with moderate-severe cognitive impairment according to MMSE scale (score 18 or lower) and/or the GDS scale (score 5 or higher)\*.
- Those with physical disability according to Barthel Index (lower to 40)
- Participants with critical acute disease who might need admission in an Intensive Care Unit (ICU).
- Life expectancy lower than six months
- Nursing home residents

<sup>\*</sup> This cut-off was selected to establish a higher sensitivity and maintain a good recruitment rate.(24)



## 7 RECRUITMENT

Participants will be recruited in Spain, United Kingdom and Italy according to legal requirements in each country. Also, we will obtain the committee approbation in the hospitals, as well as, doing a contract in each hospital. The administrative matters will be handled by CRO Business&Decision Life Sciences (Contract Research Organization).

## 7.1 INFORMED CONSENT AND ELEGIBILITY CRITERIA

Potential participants will be evaluated by authorized members of the clinical trial who will be trained to provide the necessary information to adequately explain the trial protocol and solve the issues that arise from the possible candidate to join the study team. If necessary, several members of the research team should discuss and solve the doubts concerns of the patient.

The team member will be willing to answer questions from potential participants verbally or in writing if necessary in simple, clear and understandable language. Upon acceptance by the participant, potential eligibility criteria shall be formally evaluated, if they do, he or she shall sign the informed consent (Annex 1)

The Principal Investigator (PI) will have overall responsibility for solving any problems that might arise about informed consent and supervise all study participants to ensure that everyone involved in this process are properly trained according to the ethics committee approval protocol and Guides of Good Clinical Practice (GCP) and the Declaration of Helsinki of 1996.

Informed consent will be obtained before the participant is assessed by specialists with the purposes of the study. The right of a participant to refuse to participate without giving reasons will be respected. The participant may withdraw at any time without giving reasons and without prejudice to his / her further treatment. At no time during the process of obtaining informed consent the investigator or any member of the research team coerce or influence for the patient to be part of the clinical trial.



The investigator will check if the participant has successfully completed the consent form and that it has been signed and dated correctly. The researcher must sign and date the form in the right area on the same date as the participant. The original informed consent will be filed in the archive of the researcher.

If a participant is ineligible after randomization, it shall be reported immediately to the principal investigator.

Patients who during the follow up present a moderate or severe cognitive impairment will remain in the group assigned.

## 7.2 RANDOMIZATION

After verification that the participant fulfils the eligibility criteria and signed the informed consent, allocation will be made to a control or/an intervention group.

Participants will be randomized 1:1 through the eCRF by Linkcare Company, which also will do the database.

Patient's participation in the study and the telephone number of the study contacts will always be registered in his/her clinical record.

According to the study's schedule, the intervention phase will start the sixteenth week, taking into account the adjustments of the ethics committee in each country. Follow-up will be made at hospital discharge and at the third and sixth month after discharge.

## 7.3 SAMPLE SIZE

Dependence and disability affects quality of life perception and increases health costs. Hence, this variable will be taken to calculate sample size. According to literature, the incidence of disability in frail older people is approximately 40%.

In order to avoid the estimation bias, the sample size will have at least 10 outcomes as variables. Therefore, the formula has been calculated for a 95% confidence interval to obtain at least 40 events.



$$n * p \pm z_{1-\frac{\alpha}{2}} \sqrt{n * p * (1-p)}$$

It has been assumed drop-out rate of 20% and an incidence of disability described above. Hence, the sample size should be at least 1860 participants. In each clinical setting (emergency room, general surgery, oncology, cardiology and nephrology) 310 participants should be evaluated (155 in each group: control and intervention).

In case of not obtaining the minimal sample size in each clinical setting, the pondeate models will be made. Additionally, a meta-analysis will be performed including the global effect of the intervention according to clinical setting and with a thorough sensitivity analysis.

## 7.4 STATISTICAL ANALYSIS

Firstly, subject's basal characteristics at recruitment will be analyzed. Descriptive statistics of epidemiological and clinical data will be calculated (described in section 9). This analysis will be done in a conjoint manner, according to treatment and clinical setting (emergency room, general surgery, oncology, cardiology, and nephrology).

To verify the differences between the arms of the study a Mann-Whitney test will be made. Based on the inclusion criteria, it is expected that the differences will be produced by the intervention, and not because of differences between groups.

To evaluate the intervention in each clinical setting, the effect of the intervention and its statistical significance will be determined.

These effects shall be broken down into two classes depending on the event. First the prevalence rate, and in case the event's duration could be assessed, evaluate if this duration has changed..

For each outcome described in section 4, comparisons between predictive values of the logistic models for each scale will be made in order to determine which scale is optimal in a global manner, according to clinical setting.

In case the date of death and hospitalization can be obtained, survival models will be done.



Diagram 1. Flowchart of randomized clinical trial





## 8 INTERVENTION AND CONTROL

## 8.1 CONTROL GROUP

Patients will receive medical attention according to usual medical/surgical treatment and the peculiarities of each pathology and clinical setting. In this Group of patients a Comprehensive Geriatric Assessment will be done at hospital admission and discharge. If at any case, a geriatrician consultation is required, it should be registered in the eCRF and in patient's record. The statistical analysis of these patients' data should be made, if there's enough sample throughout a sensitivity analysis.

## 8.2 INTERVENTION GROUP

Patients included in this Group will be treated by usual physician with the support of geriatrics team, who will do Comprehensive Geriatric Assessment to detect any problem in the elderly population in the clinical, functional, mental and social domains. The objective is to establish a strategy of intervention, treatment and follow-up to optimize resources and improve independency and quality of life..



## 9 ASSESMENTS DURING THE STUDY

## 9.1 BASELINE EVALUATION (visit 0= FIRST VISIT)

After the inclusion of a participant in the study, a comprehensive geriatric assessment will be done with the following parts:

**Demographics and epidemiology:**Date of birth, age, sex, race, caregiver, marital status, number of persons in the house, and, number of hospitalization in the last year, follow up by others specialist, level of education.

Medical history

Personal Medical and Surgery History should be recorded in the electronic Case Report Form (eCRF).

• Medications:

In the CRF we register all the regularly medication use (previous hospitalization)

• Functional status

Evaluate functional status with the following scales: Barthel Index, Lawton Index, measures based in performance (SPPB-Short Physical Performance Battery) and PASE Scale, Annex 2.

• Cognitive and depression:

Evaluate the results with MMSE and Geriatric Depression Scale GDS, and delirium risk with CAM scale. See Index 2.

• Physical examination:

Vital signs and physical examination as usual by the clinical investigator.

• Geriatric Syndromes Assessment:

Immobility: Falls and imbalance.

Incontinence: urinary and fecal.

Sensory deprivation

Iatrogenic: Record the numbers of falls during the hospitalization and adverse effects

Pain: assess pain using the VAS Scale. Nutritional Status:



Performed screening for nutritional status using the scale MNA (Mini Nutritional Assessment), Index 2.

• Comorbidities:

Comorbidities will be quantified by Charlson Index, Index 2.

Quality of Life:

The evaluation for the quality of life using the EuroQolfive-dimensional (EQ-5D), Index 2. Caregiver:

• Assessment for the burden of the caregiver; Will be evaluated with The Modified Caregiver Strain Scale. Index 2.

## 9.2 EVALUATION AT DISCHARGE FROM THE SPECIFIC CLINICAL SETTING

The following aspects will be assessed:

- Mortality
- Frailty assessment with L. P. Fried's scale and/or FRAIL scale. Functionality assessment with Barthel Index. Indicate the number of hospital stay in days.
- Describe if the patient change the Ward location/ medical /surgical in the hospital
   (UCI, Coronary unitetc) o )during the evolution in the hospital
- Quantification the number of test (Blood test, urine test, X- Ray, ecography, CT, etc and more specialized like: PET TAC, echocardiography, polisomnography, etc.)
- Quantification the number of consult with other specialist, social worker, paliative care. Etc.
- Usual treatment ( Register all the meditation at discharge
- Evaluate if the patient develop geriatric síndrome (page 22).
- Destination at dischargeia. (Nursing home, follow up by home care team, l HUG-GRT, day hospital, rehabilitation at home, specialist consultation, etc.)
- Evaluate the perception of the quality of life with the scale EuroQolfive-dimensional (EQ-5D).
- Burden of the caregiver with the Economics questionnaire s.
- Economics evaluation Index 3



## 9.3 EVALUATION AT 3 MONTHS OF DISCHARGE

Re-evaluate the following aspects by phone:

- Mortality
- Functionality data (Barthel index, Lawton index, PASE Scale).
- Usual medication.
- Residency at the moment.
- Frailty with the FRAIL scale..
- Data of quality of life with the scale EuroQolfive-dimensional (EQ-5D)
- Number of hospitalization and ER, indicate the cause (diagnosis)
- Caregiver burden with the economic questionaries.
- Economics evaluation, Index 3

## 9.4 EVALUATION AT 12 MONTHS OF DISCHARGE

Re-evaluate the following aspects by phone

- Mortality
- Funtionality data (Barthel index, Lawton index, PASE Scale).
- Usual medication.
- Residency at the moment.
- Frailty with the FRAIL scale. Datos de fragilidad con la escala FRAIL.
- Data of quality of life with the scale EuroQolfive-dimensional (EQ-5D)
- Number of hospitalization and ER, indicate the cause (diagnosis)
- Burden of the caregiver with the economics questionnaires.
- Economics evaluation., Index 3

## 9.5 END OF THE STUDY EVALUATION

- The study will finish at 12 months after patient's discharge with a lastphone call.
- We should make an effort to write all the data during the study, at follow up and the final evaluation.

A follow-up and investigator's tasks schedule was performed during the study. See table 2.



Table 2 Schedule of the investigation

| Intervention phase | | Initial | Discharge | | 12 month |
|---|---|---|---|---|---|
| | Eligibility&recruitment | Visit | | Follow- | Follow-up |
| | Englomity&recruitment | VISIC | | up | |
| Informed consent | X | | | | |
| | V. | *** | | | |
| Eligibility CI and CE<br>Medical history | X | X | | | |
| Usual treatment | | X | X | X | X |
| Comprehensive Geriatric | | Λ | Λ | Λ | Λ |
| Assessment | | X | | | |
| Assessment | | | | | |
| | | X | | | |
| Cognitive and depression | | ^ | | | |
| (MMSE,GDS,CAM) | | | | | |
| , | | X | | | |
| Comorbidities - Charlson I. | | Λ | X | | |
| Functional Status | | X | Λ | X | |
| | | ^ | Barthel | ^ | X |
| (Barthel I, Lawton I, PASE, | | SPBB | Dartiei | | Λ |
| SPBB) | | SPDD | | | |
| Sociodemographic data | | X | | | |
| PhysicalExam | | X | | | |
| Nutritional Status (MNA) | | X | | | |
| Permanent residence | | X | X | X | X |
| Mean hospital stay | | | X | | |
| Death | | | X | X | X |
| Frailty (Fried) | | X | X | ** | |
| Frailty(FRAIL) | | X | X | X | X |
| EuroQolfive-dimensional (EQ- | | X | X | X | X |
| 5D) | | | | | |
| Caregiver burden | | X | X | X | X |
| Relocation to other hospital | | | | | |
| services | | | X | | |
| Adverse events (iatrogenic, | | ,, | ., | | |
| falls, geriatric syndromes, etc.) | | X | X | | |
| , germanie sy mai omies, etc.) | | | | | |
| Economics evaluation | | | X | X | X |
| Checklist of complementary | | | | | |
| test during the hospitalization | | | X | | |
| test during the hospitalization | | | | | |
| Consultation to other specialist | | | v | | |
| during hospitalization | | | X | | |



| Coordination of care in different levels of care | X | | |
|--------------------------------------------------|---|---|---|
| Readmission | | X | X |
| Visits to the emergency room | | X | X |
| Nosocomial infections | X | | |

<sup>\*</sup> In case of surgical patients, who after 3 weeks since the first visit have passed and surgery hasn't been performed, evaluate the possibility of re-assessing inclusion criteria.



## 10 ECONOMIC EVALUATION

An economical evaluation of the program will be conducted to detect and handle the frail elderly in different health areas. We will conduct a comparative analysis in terms of costs and benefits of a geriatrician's intervention compared with usual care.

Information on both patients and caregivers about health resources and social services use and time spent by the caregiver will be collected. The next step is to translate this resource consumption in monetary terms. The costs will be reported in euros and in places where it is not used this coin the current exchange will take place.

The total cost is the sum of three different types of costs: directly derivate from care; formal care costs (professional) and informal care costs (family and friends)

## Direct health care costs:

These costs are related to inpatient treatment, outpatient treatment, medicines, etc. These are estimated from the use of health services by assigning a monetary value for each resource used.

Health resources will be identified and measured through questionnaires. Each center will give us the price or the monetary value of each resource. If some of this information is not available, it will be obtained from a systematic review of studies of cost of illness for each country.

### Formal care costs (Social Services):

Formal care includes those generated by social services which can be public or privately funded institutions such as day care centers, remote assistance, scheduled home care, etc. These costs will be identified, measured and evaluated through questionnaires. Ideally, members of each research team from each center must provide to the economic team price and monetary values (unit costs) of resources for social services.

If data about unit cost of social services are not available, a review of the literature will be performed to obtain the data by country.



## Social costs (informal care)

Informal care includes different types of unpaid support which serve to compensate for the inability of subjects, usually provided by relatives or friends. This information is obtained from questionnaires applied directly to caregivers in which time spent on helping the elderly in basic Activities of Daily Living and Instrumental Activities will be specified. The time spent on these activities will be evaluated in monetary terms using 'proxy goodmethod "or" replacement method "which assesses the time spent on informal care adjusted to market prices of a professional who has to do this work (social service Careful formal).

The economic evaluation will be developed to take into account several aspects: financing health care (including only direct health costs), finance formal care (including the direct costs of health and social services) and social perspective (including all relevant costs: direct medical care + formal care (social services) and informal care.

### **Outcome measures:**

## Cost-effectiveness analysis

The cost-effectiveness analysis (CEA) is the most common test used in health economics to decide between different treatments for the same condition. In a CEA, the costs are measured in monetary units, while the benefits are measured as outcomes or in natural units. "Incremental cost-effectiveness ratio" (ICER) is estimated to show a difference in health outcomes per unit cost, after a follow-up period between intervention and usual care. The incremental cost-effectiveness is expressed by the following relation:

$$ICER = \frac{C_a - C_b}{B_a - B_b}$$

Where Ca is the cost of the intervention group and Cb is the cost of the usual care group. Ba will be health benefits in the intervention group and Bb health benefits in the usual care group, both measured in terms of change of the clinical results of the baseline.

In this study the primary outcomes will be the difference in functional status after the intervention compared with usual care group. This study will assess the cost-effectiveness of the intervention of a geriatrician compared with usual care from the perspective of society and the health care system.



Complementing the main cost-effectiveness analysis, we will develop several parallel cost effectiveness analysis to the extent that effective change. The results that we will use are: hospitalization rate and readmission, lenght of hospitalization and in the Emergency department, episodes of delirium and nosocomial infection, post-surgical complications as a whole and by surgical procedure, number of inappropriate drugs, adherence to treatment, permanent institutionalization rate, survival rate, preventable side effects due to under / over / mismanagement on caregiver burden.

## **Cost-utility analysis:**

Cost-utility analysis (ACU] is an evolution of cost-effectiveness analysis, in which the interference effects are measured in a unit that synthesizes the lifespan and quality of life. The best and better known measure is the quality of life-adjusted per quality (QALY QALY or in its Anglo-Saxon sense). The QALYs are calculated by weighting the survival time (years of age) with quality adjustment thereof, called utility, which represents the preference values in relation to different health states (reference). For the purpose, the EQ-5D-5L instrument will be used. The incremental cost-utility relation answers the following expression:

ACUincremental = (Ca - Cb) / (AVAC(a) - AVAC(b))

## **Statistical analysis:**

A descriptive analysis of the main resources used in health care, social services and informal care will be performed.

This includes basic statistics such as means, medians, standard deviations, skewness, kurtosis, ranges, bivariate analysis using different cost elements and individual characteristics (sex, age,...) and health outcomes.

Because different distributions are expected from major cost components, we hope to develop different multivariate estimation methods. As we expect a non-normal distribution of the estimated costs, an alternative analysis would be the use of GLM models grouped by clusters, where depending on the distribution of the estimated costs (distribution Gamma, Poisson or Gaussian), will be used the most suitable method of empirical analysis. Another alternative, if the necessary information is obtained, could be an analysis using multilevel models of 2 or 3 grade (Recital country and center). The costs



of health care could also be analyzed by a normal multivariate model (clustering) or lognormal and the ordinary least square regression will be used to estimate the determinants of health care costs. In contrast, for the analysis of formal and informal care costs, we expect to use simple probit or ordered probit models, whether formal and informal care for a large number of people in the study is provided.



## 11. APPENDIX

## **APPENDIX 1**

## STUDY TITLE:

# FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFERRENT CLINICAL SETTINGS

(Intervention phase).

## SUBJECT'S INFORMATION FORM

Sponsor: FUNDACIÓN PARA INVESTIGACIÓN BIOMÉDICA DEL HOSPITAL UNIVERSITARIO DE GETAFE

Project leader: Prof. Leocadio Rodríguez Mañas



## **SUBJECT INFORMATION FORM**

**Study Title:** FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFFERENT CLINICAL SETTINGS

Investigator: Prof. Leocadio Rodríguez Mañas. Hospital de Getafe.

## What is this study about? What are the outcomes?

You are invited to participate in a research study because you are somebody who can meet the clinical criteria for frailty syndrome.

This syndrome (frailty) includes criteria such as: weakness, weight loss, walking speed, among others. This syndrome is associated with higher risk of developing dependency and disability. Your physician has checked that you meet the criteria for diagnosis of this syndrome.

In this study we evaluate the usefulness of a screening program of frail subjects using certain scales, and measure the benefit that suppose to the subject to associate the intervention of a geriatrician to usual clinical practice. In this study we will not test the efficacy of any new drug.

The aim of this study is to assess whether, through the intervention of a geriatrician can change the course of frailty and reduce the occurrence of adverse events from the health point of view.

A total of 1500 subjects are estimated to participate in 6 hospitals distributed by three European countries. The study was approved by the Ethics Committee of the Hospital Universitario de Getafe and ethics committees of the participating centers. It is also approved by the competent bodies of the regions concerned. It will be executed following the Declaration of Helsinki and the requirements of the Law 14/2007 of Biomedical Research. The study will last for three years.



## How this study was done?

Each hospital will select a group of approximately 250 individuals who meet the criteria to participate in the study. These people will be informed about the study and asked, if they agree to participate, to sign this informed consent form. Once subjects are selected through a randomized system (similar to throwing a coin), it is determined in which study group will participate. Half of the patients selected will participate in usual clinical practice group (control group) and half the group will receive care from a geriatrician (intervention group).

**If you belong to the control group**, will follow the recommendations, actions and treatment indicated for your specialist doctor. Nothing will change of normal medical practice.

Still, in order to assess the results of usual medical action a geriatrician will hold a series of questions when hospitalization, and following in three months and one year (the latter two are made by telephone calls).

If you are allocated to the intervention group: you will be followed by your corresponding specialist as in usual clinical practice and by a geriatrician. The geriatrician will take into account his medical criteria, always with the consent if the rest of the physicians treating you. The geriatrician will make questions about your physical, mental, social and nutritional state.

Follow-up will be made after discharge at 3 month and at 12 month (by telephone call).

What are the potential benefits and risks associated to the study? You must know this study will be supervised by experienced health professionals as doctors and nurses. It is possible that you will not obtain any benefit for the study and you can even experience some secondary effect associated to any treatment or complementary test. Some of the information obtained in this study may help improve elders quality of life, improve the capacity of doing activities of daily living or avoiding institutionalization in some cases..



## Your participation is voluntary

I you want to participate in this study, once you have read and understood this information form, and all of your questions have been answered, you must communicate your decision to your physician. You are free to abandon the study at any time without giving any explanations, and this will not change the relationship with your physician. Your physician could retire you from the study if you do not follow the given instructions or because he/she considers it will benefit your health status or on the assumption the study is cancelled. If this occurred, you will be informed the reason of its ending.

Data collected at the moment of your abandonment will be used for the objectives originally foreseen.

## Review of the original documents, confidentiality and personal data protection.

With the aim to guarantee feasibility of the collected data, the designated personal by the promoter, and eventually the health authorities and/or members of the Investigation Ethics Committee, will be allowed to access clinical records of the subject where you will be identified as main caregiver, always respecting confidentiality. Treatment, communication, and personal data transfer of every participating subject in this study will be adjusted to what is established in the Law 15/1999 of Personal Data Protection.

Data collected in the study will be identified by a numeric code and just the study physician and collaborators will be able to connect that data to you.

Any additional information that could be identifiable will be kept and processed in a secure way by informatical media by the promoter or the company designated by him/her.

Data could be transferred to other countries or collaborative groups in the study as long as they apply the necessary measures to protect personal information, transferring them in a coded way.

() frailclinic

You can exercise your right, according to current legislation, of rectifying,

cancelling o opposing, according to your personal data, talking directly to your

study physician.

**Results publication** 

The study results will be communicated to the scientific community through

congresses and/or publications. In any way, there will be no information that could

identify you in these publications.

If during the study, any relevant information that could be useful to you emerges, it

will be communicated through your study physician.

Additional information

The study meets the current Spanish legislations(Law 14/2007 of Biomedical

Investigation). According to the Spanish legislation, the promoter commits to

subscribe to an insurance policy before the beginning of the study to cover for

adverse events that could be produced during the study.

The patient should know that he/she will not receive any economic compensation

or reimbursement of expenses due to its participation in the study.

This study is financed by the CE "HEALTH-2013" PROJECTS.

You can discuss any of the information given with your attending, family or friends

before taking any decision concerning your participation in the study. If you have

any doubt or any event arises during the study, you can talk to:

Name of the Investigation Clinician: Mónica Ballesteros.

Address: Carretera de Toledo, km 12,500, 28905 Getafe, Madrid

Phone number: +34 916839360 ext. 2760

You will be given a copy of this document with date and signature.

34



## Study Title:

## FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFFERENT CLINICAL SETTINGS. INTERVENTION PHASE.

| I, (Name and Last Na | me) |
|---|---|
| Have read the information form I've l | oeen given. |
| I have been able to ask questions abo | ut the study. |
| I have received enough information a (Name of the Investigator) | about the study. I have talked to: |
| I understand that my participation if the study willingly: $1^{\circ}$ . Whenever I wa | s voluntary. I understand that I can abandor<br>nt. |
| 2º.Without giving any explication. | |
| 3º.It will not change in any way my participate in the study. SUBJECT: | plan of care. I willingly give my consent to |
| Signature: | Date |
| Name | |
| INVESTIGATOR Signature: | Date |
| Name | |
| WITNESS (if needed): | |
| Signature | Date Name: |



## STUDY TITLE:

## FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFFERENT CLINICAL SETTINGS (Intervention Phase)

## INFORMATION FORM FOR PRINCIPAL CAREGIVER

Sponsor: FUNDACIÓN PARA INVESTIGACION BIOMÉDICA
DEL HOSPITAL UNIVERSITARIO DE GETAFE

Leader of the Project: Prof. Leocadio Rodríguez Mañas


#### INFORMATION FORM FOR THE MAIN CAREGIVER

**Study Title:**:FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFFERENT CLINICAL SETTINGS.

Investigator: Prof. Leocadio Rodríguez Mañas. Hospital Getafe

#### What is the study about? What are the objectives?

You are being invited to participate in an investigation Project because you are the main caregiver of a person who can meet clinical criteria of Frailty. You are the main caregiver because you are the one that helps him/her the most with Activities of Daily Living, or the one who is asked the most for help and is not hired for it.

Frailty has different criteria as: weakness, weight loss, gait speed, among others. This syndrome is associated to a higher risk of dependency and disability. In this study we want to evaluate the usefulness of a program to detect frailty, with the use of determined scales, as to assess the benefits the subject obtains with associating a geriatrician's intervention to the usual clinical practice. This study is not aimed to prove the efficacy of any new medication..

The study's objective is to evaluate if the evolution of frailty and reduction of adverse events from the medical point of view can be changed through a geriatrician's intervention.

1500 subjects are estimated to participate in all 6 hospitals distributed in 3 European countries. The study is approved by the Ethics Committee of the Hospital Universitario de Getafe and ethics committees in all of the other participating centers. It is also approved by the competent organs of the implied communities. It is going to be made following the Helsinki Declaration and the demands established by the Law 14/2007 of Biomedical Investigation. The study has a three years duration.



#### What is my participation about?

Each health center will choose a group of 200 subjects who meet the participation criteria. These subjects will be asked to identify their main caregiver, if applicable. You, as caregiver, will be asked to answer two different polls about the subject's care. They will be done three times; during hospitalization, at three month and at the first year of follow-up, the latest by telephone call.

Which are the potential benefits and risks associated to the study? Participating in this study will not imply any benefit or risk because we are only asking you to fill questionnaires that will take some of your time. Obtained information in the study could help to improve quality of life of elders, improving their capacity to do certain activities or avoiding institutionalization in some cases.

#### Your participation is voluntary

If you want to participate in this study, once you have read and understood this information form, and all of your questions have been answered, you must communicate your decision to your physician. You are free to abandon the study at any time without giving any explanations, and this will not change the relationship with your physician. Your physician could retire you from the study if you do not follow the given instructions or because he/she considers it will benefit your health status or on the assumption the study is cancelled. If this occurred, you will be informed the reason of its ending.

Data collected at the moment of your abandonment will be used for the objectives originally foreseen.

## Review of the original documents, confidentiality and personal data protection.

With the aim to guarantee feasibility of the collected data, the designated personel by the promoter, and eventually the health authorities and/or members of the Investigation Ethics Committee, will be allowed to access clinical records of the subject where you will be identified as main caregiver, always respecting



confidentiality. Treatment, communication, and personal data transferof every participating subject in this study will be adjusted to what is established in the Law 15/1999 of Personal Data Protection.

Data collected in the study will be identified by a numeric code and just the study physician and collaborators will be able to connect that data to you. Any aditional information that could be identifiable will be kept and processed in a secure way by informatical media by the promoter or the company designated by him/her. Data could be transferred to other countries or collaborative groups in the study as long as they apply the necessary measures to protect personal information, transferring them in a coded way.

You can exercise your right, according to current legislation, of rectifying, cancelling o opposing, according to your personal data, talking directly to your study physician.

#### **Results publication**

The study results will be communicated to the scientific community through congresses and/or publications. In any way, there will be no information that could identify you in these publications. If during the study, any relevant information that could be useful to you emerges, it will be communicated through your study physician.

**Additional information:** The present study follows current Spanish legislation (Law 14/2007 of Biomedical Investigation). According to Spanish legislation, the promoter compromises to subscribe an insurance policy before the beginning of the study that covers for adverse events that could emerge during the study. You should know that you will not receive any economical compensation or reimbursement for any of the expenses associated to your participation in the study. This study is financed by the CE "HEALTH-2013" PROJECTS.

You can comment the information received with your physician, family or friends before making any decision concerning your participation in the study. Name of the study physician: Mónica Ballesteros



Address: Carretera de Toledo, km 12,500, 28905 Getafe, Madrid

Phone number: +34 916839360 extension 2760

You will receive a copy of this document with date and signature. Study title: Feasibility and Effectiveness of the Implementation of Programs to Screen and Manage Frail Older Patients in different clinical settings.



## Study Title

# FEASIBILITY AND EFFECTIVENESS OF THE IMPLEMENTATION OF PROGRAMS TO SCREEN AND MANAGE FRAIL OLDER PATIENTS IN DIFFERENT CLINICAL SETTINGS. INTERVENTION PHASE.

| I, (Name and Last N | ame) |
|---|---|
| Have read the information form I've | e been given. |
| I have been able to ask questions ab | oout the study. |
| I have received enough information (Name of the Investigator) | about the study. I have talked to: |
| I understand that my participation the study willingly: $1^{\circ}$ . Whenever I v | is voluntary .I understand that I can abandon<br>vant. |
| 2º.Without giving any explication. | |
| 3º.It will not change in any way n<br>participate in the study. SUBJECT: | ny plan of care. I willingly give my consent to |
| Signature: | Date |
| Name | |
| Investigator's Signature : | Date |
| Name | |
| WITNESS (if needed): | |
| Signature | DateName: |



#### **APPENDIX 2**

#### FRIED'S CRITERIA

#### 1- Weight loss:

We have to ask the patient if he or she has lost weight unintentionally in the past year, and if the loss was greater than 4,5 kg (10 lb).

- > YES (1)
- > NO (0)

#### 2- Exhaustion:

- "I felt that everything I did was an effort during the past week"
- I could not get "going"

If SOME (OR BOTH) answers are YES, one point for frailty will be counted.

#### 3- Physical activity:

Does the patient perform less than or equal to the physical activity indicated weekly?

Men:  $< 383 \text{ kcal / week (walking } \le 2 \text{ hours and } 30 \text{ minutes / week)}$ 

Women: < 270 kcal / week (walking < 2 hours / week)

We ask the patient to respond with YES or NO if he/she performs these activities.

If they answer YES, one point for frailty will be counted.

4- *Slowness:* measured as the time it takes for the patient to travel 15 feet to their usual walking speed.

| SEX | Height(CM) | CUT OFF |
|-------|------------|----------------|
| MEN | ≤173 cm | <u>≥</u> 7s |
| | >173 cm | <u>&gt;</u> 6s |
| WOMEN | ≤159 cm | <u>≥</u> 7s |
| | >159 cm | <u>≥</u> 6s |

This is done as follows: we will indicate to the patient to stand immediately behind the starting line, we will tell him/her to start walking "as he/she usually does". The patient is then stopped. We will do the test twice and we will take the best score of the two. The time will be recorded in seconds.

5- **Weakness:** Assessed by grip strength.

| BMI♂ | CUT-OFF | BMI♀ | CUT-OFF |
|---------|---------|---------|---------|
| ≤24 | <29kg | ≤23 | <17kg |
| 24,1-26 | <30kg | 23,1-26 | <17,3kg |
| 26,1-28 | <30kg | 26,1-29 | <18kg |
| > 28 | <32kg | >29 | <21 kg |



He/she will rest for about 30 seconds, and he/she will repeat the exercise two more times. We will record the best of all results.



#### **FRAIL**

- 1.- <u>Fatigue</u> is measured by asking respondents how much time during the past 4 weeks they have felt tired with responses of "all of the time" or "most of the time" scored as 1 point.
- 2.- **Resistance** is assessed by asking participants if they have had any difficulty walking up 10 steps alone without resting and without aids.
- 3.- **Ambulation** is assessed by asking if they had any difficulty walking several hundred meters alone and without aids: a yes response is scored as 1 point.
- 4.- <u>Illness</u> is scored 1 for respondents who report 5 or more illnesses out of 11 total illnesses:(hypertension, diabetes, cancer (other than a minor skin cancer), chronic lung disease, heart attack, congestive heart failure, angina, asthma, arthritis, stroke, and kidney disease).
- 5.- **Loss of weight** is scored 1 for respondents with a weight decline of 5 % or greater within the past 12 months based on self-report.



### **EUROQL 5D 5L:( (25)**

Under each heading, please tick the ONE box that best describes your health TODAY

| MOBILITY |
|---|
| I have no problems in walking about |
| I have slight problems in walking about |
| I have moderate problems in walking about |
| I have severe problems in walking about |
| I am unable to walk about |
| SELF-CARE |
| I have no problems washing or dressing myself |
| I have slight problems washing or dressing myself |
| I have moderate problems washing or dressing myself |
| I have severe problems washing or dressing myself |
| I am unable to wash or dress myself |
| <b>USUAL ACTIVITIES</b> (e.g. work, study, housework, family or leisure activities) |
| I have no problems doing my usual activities |
| I have slight problems doing my usual activities |
| I have moderate problems doing my usual activities |
| I have severe problems doing my usual activities |
| I am unable to do my usual activities |
| PAIN / DISCOMFORT |
| I have no pain or discomfort |
| I have slight pain or discomfort |
| I have moderate pain or discomfort |
| I have severe pain or discomfort |
| I have extreme pain or discomfort |
| ANXIETY / DEPRESSION |
| I am not anxious or depressed |
| I am slightly anxious or depressed |
| I am moderately anxious or depressed |
| I am severely anxious or depressed |
| I am extremely anxious or depressed |



 We would like to know how good or bad your health is TODAY.

- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
  0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.
  - YOUR HEALTH TODAY =

The best health you can imagine



The worst health you can imagine



## **Barthel Index (Basic activities of daily living)**

| Feeding | | |
|---|---|---|
| 0 = unable | | |
| 5 = needs help cutting, spreading butter, etc., or requires | | F 10 |
| modified diet | 0 | 5 10 |
| 10 = independent | | |
| • | | |
| Bathing | | |
| 0 = dependent | | 5 |
| 5 = independent (or in shower) | | 3 |
| Grooming | | |
| 0 = needs to help with personal care | | |
| 5 = independent face/hair/teeth/shaving (implements | | _ |
| provided) | 0 | 5 |
| Dressing | | |
| 0 = dependent | | |
| 5 = needs help but can do about half unaided | | |
| 10 = independent (including buttons, zips, laces) | 0 | 5 10 |
| Bowels | | |
| 0 = incontinent (or needs to be given enemas) | <b> </b> | |
| , , | | |
| 5 = occasionalaccident | 0 | 5 10 |
| 10 = continent | | |
| Bladder | | |
| 0 = incontinent, or catheterized and unable to manage | | |
| alone | 0 | 5 10 |
| 5 = occasionalaccident | | |
| 10 = continent | | |
| Toilet Use | | |
| 0 = dependent | | |
| 5 = needs help, but can do something alone | | |
| 10 = independent (on and off, dressing, wiping) | 0 | 5 10 |
| Transfers (bed to chair and back) | | |
| 0 = unable, no sitting balance | | 5 10 15 |
| 5 = major help (one/two people,physical), can sit | | 3 10 13 |
| 10 = minor help (verbal or physical) | | |
| 15 = independent | | |
| Mobility (on level surfaces) | | |
| 0 = immobile or < 50 yards | | |
| 5 = wheelchair independent (inc.corners)>50 yds | | |
| 10 = walks with help of one person (verbal or physical) > | | |
| 50 yards | 0 | 5 10 15 |
| 15 = independent (but may use any aid; for example, | | |
| stick) > 50 yards | | |
| Stairs | | |
| 0 = unable | <sub> </sub> | |
| 5 = needs help (verbal, physical, carrying aid) | 0 | 5 10 |
| 10 = independent | | |
| TOTAL (0-100) | | |
| 1111 / 4 111-111111 | | |



## THE LAWTON INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE

| A. Ability to Use Telephone | E. Laundry |
|---|---|
| 1. Operates telephone on own initiative; looks up | 1. Does personal laundry completely |
| and dials numbers1 | 2. Launders small items, rinses socks, stockings, etc1 |
| 2. Dials a few well-known numbers1 | 3. All laundry must be done by others0 |
| 3. Answers telephone, but does not dial1 | |
| 4. Does not use telephone at all0 | |
| | F. Mode of Transportation |
| | 1. Travels independently on public transportation |
| B. Shopping | or drives own car1 |
| 1. Takes care of all shopping needs independently1 | 2. Arranges own travel via taxi, but does not |
| 2. Shops independently for small purchases0 | otherwise use public transportation1 |
| 3. Needs to be accompanied on any shopping trip0 | 3. Travels on public transportation when assisted |
| 4. Completely unable to shop0 | or accompanied by another1 |
| | 4. Travel limited to taxi or automobile with |
| | assistance of another |
| C. Food Preparation | 5. Does not travel at all0 |
| 1. Plans, prepares, and serves adequate | |
| meals independently1 | C. Doomoneihilitu fou Ouun Medientiene |
| 2. Prepares adequate meals if supplied | G. Responsibility for Own Medications |
| with ingredients0 | Is responsible for taking medication in correct |
| 3. Heats and serves prepared meals or prepares meals | dosages at correct time |
| but does not maintain adequate diet | Takes responsibility if medication is prepared in advance in separate dosages |
| 4. Needs to have meals prepared and served0 | 3. Is not capable of dispensing own medication0 |
| | 5. Is not capable of dispensing own medication |
| D. Housekeeping | |
| 1. Maintains house alone with occasion assistance | H. Ability to Handle Finances |
| (heavy work)1 | 1. Manages financial matters independently (budgets, |
| 2. Performs light daily tasks such as dishwashing, | writes checks, pays rent and bills, goes to bank); |
| bed making1 | collects and keeps track of income1 |
| 3. Performs light daily tasks, but cannot maintain | 2. Manages day-to-day purchases, but needs help |
| acceptable level of cleanliness1 | with banking, major purchases, etc1 |
| 4. Needs help with all home maintenance tasks1 | 3. Incapable of handling money0 |
| 5. Does not participate in any housekeeping tasks0 | |



#### **GERIATRIC DEPRESSION SCALE (GDS)**

Choose the best answer for how you have felt over the past week:

1. Are you basically satisfied with your life?

YES / NO

2. Have you dropped many of your activities and interests?

YES / NO

3. Do you feel that your life is empty?

YES / NO

4. Do you often get bored?

YES / NO

5. Are you in good spirits most of the time?

YES / NO

6. Are you afraid that something bad is going to happen to you?

YES / NO

7. Do you feel happy most of the time?

YES / NO

8. Do you often feel helpless?

YES / NO

9. Do you prefer to stay at home, rather than going out and doing new things?

YES / NO

10. Do you feel you have more problems with memory than most?

YES / NO

11. Do you think it is wonderful to be alive now?

YES / NO

12. Do you feel pretty worthless the way you are now?

YES / NO

13. Do you feel full of energy?

YES / NO

14. Do you feel that your situation is hopeless?

YES / NO

15. Do you think that most people are better off than you are?

YES / NO



#### **CAREGIVER BURDEN:**

#### **MODIFIED CAREGIVER STRAIN SCALE (CSS)**

Being available to help or regularly caring for someone can be difficult and disruptive. Which of the following statements apply to you...? We have included some examples that are common caregiver experiences to help you think about each item. Your situation may be slightly different, but the item could still apply. For each statement, please circle <u>one</u> answer (Not at all; Sometimes; Often; or

Always) as appropriate.

| | | onvenient (e.g. becaus<br>it's a long drive over t | | erson takes so much |
|---|---|---|---|---|
| Not at | all | Sometimes | Often | Always |
| 2. | - | o is disturbed (e.g. bed<br>and out of bed, or wa | - | on I care for needs help at night). |
| Not at | all | Sometimes | Often | Always |
| 3. | | nysical strain (e.g. beca<br>l tasks for which effor | | |
| | P | | | |
| Not at | • | Sometimes | Often | Always |
| | all | fining (e.g. because th | | Always icts free time or cannot |
| | It is congo visiti | fining (e.g. because th | | |
| 4. | It is congo visiti | fining (e.g. because the | e person restri | icts free time or cannot |
| 4. | It is congo visiti | fining (e.g. because th<br>ng). <b>Sometimes</b> | e person restri Often tments (e.g. be | icts free time or cannot Always cause helping the perso |

job; could not go on holiday).

**Sometimes** 

**Often** 

**Always** 

Not at all

50



7. There have been other demands on my time (e.g. from other family members). Not at all **Sometimes** Often **Always** 8. There have been emotional adjustments (e.g. because of arguments with the person). Not at all **Sometimes Often Always** 9. Some behaviour is upsetting (e.g. because of incontinence: or he or she resists help). Not at all **Sometimes** Always **Often** 10. It is upsetting to find the person has changed from their former self (e.g. they are so different from before). Not at all **Sometimes** Often Always 11. There have been work adjustments (e.g. because of having to take time off caring for the person). Not at all **Sometimes Often Always** 12. It is a financial strain Not at all **Sometimes Often Always** 13. I am feeling completely overwhelmed (e.g. because of worry about the person; concerns about how I will manage). Not at all Sometimes Often Always THANK YOU FOR YOUR TIME AND HELP



## RISK OF DELIRIUM - CAM(Confusion Assessment Method)

| Table 1<br>CAM-ICU Features and Descriptions <sup>6</sup> | | | |
|---|---|---|---|
| 1. Acute Onset or Fluctuating Course | | <u>Absent</u> | <u>Present</u> |
| Is there evidence of an acute change in mental state | us from baseline? | | |
| or | | | |
| Did the (abnormal) behavior fluctuate during the paincrease and decrease in severity as evidenced by flu<br>GCS, or previous delirium assessment? | | | |
| 2. <u>Inattention</u> | | <u>Absent</u> | <u>Present</u> |
| Did the patient have difficulty focusing attention as evid<br>or visual component of the ASE? | denced by scores <8 on either the auditory | | |
| 3. <u>Disorganized Thinking</u> | | <u>Absent</u> | <u>Present</u> |
| Is there evidence of disorganized or incoherent thinking of the 4 questions and/or inability to follow the comma | | | |
| Questions (Alternate Set A and Set B): | | | |
| Set A | Set B | | |
| 1. Will a stone float on water? | <ol> <li>Will a leaf float on water?</li> </ol> | | |
| 2. Are there fish in the sea? | 2. Are there elephants in the sea? | | |
| 3. Does 1 pound weigh more than 2 pounds? | 3. Do 2 pounds weigh more than 1 po | ound? | |
| 4. Can you use a hammer to pound a nail? | 4. Can you use a hammer to cut woo | od? | |
| Other: | | | |
| <ol> <li>Are you having any unclear thinking?</li> </ol> | | | |
| 2. Hold up this many fingers (examiner holds two f | ingers in front of patient). | | |
| 3. Now do the same thing with the other hand (no | ot repeating the number of fingers). | | |
| 4. Altered Level of Consciousness | | <u>Absent</u> | <u>Present</u> |
| Is the patient's level of consciousness anything other or stupor (eg, RASS other than "0" at time of assessment | | | |
| Overall CAM-ICU: | | <u>Yes</u> | No |
| Features 1 and 2 and either Feature 3 or 4 | | | |
| CAM-ICU=Confusion Assessment Method for the Intensive Care Unit<br>Screening Examination. | t; RASS=Richmond Agitation-Sedation Scale; GCS=Gk | asgow Coma Sc | ale; ASE=Attentic |

Pun BT, Ely EW. Primary Psychiatry. Vol 11, No 11. 2004.

52



#### **SPPB (SHORT PHYSICAL PERFORMANCE BATTERY)**





#### PHYSICAL ACTIVITY SCALE FOR THE ELDERLY (PASE)

### **INSTRUCTIONS:**

Please complete this questionnaire by either circling the correct response or filling in the blank. Here is an example:

During the past 7 days, how often have you seen the sun?

Answer all items as accurately as possible. All information is strictly confidential.



#### LEISURE TIME ACTIVITY

1.

| [0.] NEVER<br><b>↓</b> | [1.] SELDOM<br>(1-2 DAYS) | [2.] SOMETIMES<br>(3-4 DAYS) | [3.] OFTEN<br>(5-7 DAYS) |
|---|---|---|---|
| GO TO Q.#2 | • | • | ₩ ′ |
| la. | What were these acti | vities? | |
| 1b. | A CONTRACTOR OF THE CONTRACTOR CONTRACTOR | ny hours per day did | you engage in these |
| 1b. | sitting activities? | | |
| 1b. | sitting activities? | ny hours per day did UR [2.] 1 BUT LESS 7 | |

Over the past 7 days, how often did you participate in sitting activities such as reading,

2. Over the past 7 days, how often did you take a walk outside your home or yard for any reason? For example, for fun or exercise, walking to work, walking the dog, etc.?





| 3. | Over the past 7 days, how often did you engage in light sport or recreational activities such as bowling, golf with a cart, shuffleboard, fishing from a boat or pier or other similar activities? | | | | | Ø. | |
|---|---|---|---|---|---|---|---|
| | [0.] NEVER | | [1.] SELDOM<br>(1-2 DAYS)<br><b>↓</b> | [2.] | SOMETIMES (3-4 DAYS) ◆ | [3.] OFTEN (5-7 DAYS) <b>▼</b> | |
| | | 3a. | What were these a | ctiviti | es? | | |
| | | 3b. | On average, how n<br>light sport or recre | 10 | | l you engage in these | |
| | | | [1.] LESS THAN 1 F | HOUR | [2.] 1 BUT LESS | THAN 2 HOURS | |
| | | | [3.] 2-4 HOURS | | [4.] MORE THA | N 4 HOURS | |
| 4. | activities s | uch as<br>all or ot | 5 2 | room c | No. of the second secon | e sport and recreational<br>, ice skating, golf without<br>[3.] OFTEN<br>(5-7 DAYS) | a |
| | GO TO Q.#5 | t.<br>H | (1-2 DA 15)<br>• | | (3-4 DA13)<br><b>↓</b> | (3-7 DAYS) | |
| | 4a. What were these activities? | | | | | | |
| | 4b. On average, how many hours per day did you engage in these moderate sport and recreational activities? | | | | | | |

[1.] LESS THAN 1 HOUR [2.] 1 BUT LESS THAN 2 HOURS

[4.] MORE THAN 4 HOURS

[3.] 2-4 HOURS



| 5. | Over the past 7 days, how often did you engage in strenuous sport and recreational activities such as jogging, swimming, cycling, singles tennis, aerobic dance, skiing (downhill or cross-country) or other similar activities? | | | | |
|---|---|---|---|---|---|
| | [0.] NEVER<br><b>↓</b> GO TO Q.#6 | | [1.] SELDOM (1-2 DAYS) | [2.] SOMETIMES (3-4 DAYS) | [3.] OFTEN<br>(5-7 DAYS) |
| | GO 10 Q.#0 | | • | • | • |
| | 5 | 5a. | What were these activ | vities? | |
| | 5 | 5b. | On average, how man strenuous sport and re | | |
| | | | [1.] LESS THAN 1 HOU | UR [2.] 1 BUT LESS T | HAN 2 HOURS |
| | | | [3.] 2-4 HOURS | [4.] MORE THAN | 4 HOURS |
| 6. | 10 Table 1 | | nys, how often did you<br>arance, such as lifting w | | eifically to increase muscle c.? |
| | [0.] NEVER | | [1.] SELDOM | [2.] SOMETIMES | [3.] OFTEN |
| | <b>↓</b><br>GO TO Q.#7 | | (1-2 DAYS)<br><b>↓</b> | (3-4 DAYS) | (5-7 DAYS)<br><b>Ψ</b> |
| | 6 | ба. | What were these activities? | | |
| | | 6b.<br>increa | On average, how many hours per day did you engage in exercises to ase muscle strength and endurance? | | |
| | | | [1.] LESS THAN 1 HOU | JR [2.] 1 BUT LESS T | HAN 2 HOURS |
| | | | [3.] 2-4 HOURS | [4.] MORE THAN | 4 HOURS |



## HOUSEHOLD ACTIVITY

| 7. | | During the past 7 days, have you done any light housework, such as dusting washing dishes? | | |
|---|---|---|---|---|
| | [1.] No | O [2.] YES | | |
| 8. | | g the past 7 days, have you done any heavy ho<br>ming, scrubbing floors, washing windows, or o | | |
| | [1.] No | O [2.] YES | | |
| 9. | Durin | During the past 7 days, did you engage in any of the following activities? | | |
| | | Please answer <u>YES</u> or <u>NO</u> for each item. | | |
| | a. | Home repairs like painting, | <u>NO</u> | YES |
| | | wallpapering, electrical work, etc. | 1 | 2 |
| | b. | Lawn work or yard care, including snow or leaf removal, wood chopping, etc. | 1 | 2 |
| | c. | Outdoor gardening | 1 | 2 |
| | d. | Caring for an other person. | | |

such as children, dependent

spouse, or an other adult

2

1



## WORK-RELATED ACTIVITY

| 10. | During the p | oast 7 days. | , did you | work for p | oay or as a v | olunteer? |
|---|---|---|---|---|---|---|

[1.] NO [2.] YES

| 10a.<br>and/o | How many hours per week did you work for pay r as a volunteer? HOURS |
|---|---|
| | Which of the following categories best describes mount of physical activity required on your job r volunteer work? |
| [1] | Mainly sitting with slight arm movements. [Examples: office worker, watchmaker, seated assembly line worker, bus driver, etc.] |
| [2] | Sitting or standing with some walking. [Examples: cashier, general office worker, light tool and machinery worker.] |
| [3] | Walking, with some handling of materials generally weighing less than 50 pounds. [Examples: mailman, waiter/waitress, construction worker, heavy tool and machinery worker.] |
| [4] | Walking and heavy manual work often requiring handling of materials weighing over 50 pounds. [Examples: lumberjack, stone mason, farm or general laborer.] |



#### **NUTRITIONAL ASSESMENT:**

© Nestlé, 1994, Revision 2009. N67200 12/99 10M For more information: www.mna-elderly.com

## Mini Nutritional Assessment MNA®

## Nestlé Nutrition(nstitute

| Last name: | | First name: | |
|---|---|---|---|
| Sex: Age: | Weight, kg: | Height, cm: | Date: |
| Complete the screen by filling in the boxes with the Add the numbers for the screen. If score is 11 or le | | sessment to gain a Malnutrition Indicator Sco | ore. |
| Screening | | J How many full meals does the pat | ient eat daily? |
| A Has food intake declined over the past 3 m of appetite, digestive problems, chewing or difficulties? | | 0 = 1 meal<br>1 = 2 meals<br>2 = 3 meals | |
| 0 = severe decrease in food intake 1 = moderate decrease in food intake 2 = no decrease in food intake | | K Selected consumption markers fo At least one serving of dairy product (milk, cheese, yoghurt) per day Two or more servings of legumes | • |
| B Weight loss during the last 3 months 0 = weight loss greater than 3kg (6.6lbs) 1 = does not know 2 = weight loss between 1 and 3kg (2.2 and 6. | 6 lbs) | or eggs per week • Meat, fish or poultry every day 0.0 = if 0 or 1 yes 0.5 = if 2 yes 1.0 = if 3 yes | yes 🗌 no 🗍 |
| 3 = no weight loss | | L Consumes two or more servings | of fruit or vegetables |
| C Mobility 0 = bed or chair bound 1 = able to get out of bed / chair but does not of | io out | <b>per day?</b><br>0 = no 1 = yes | |
| 2 = goes out | | M How much fluid (water, juice, coff consumed per day? | ee, tea, milk) is |
| D Has suffered psychological stress or acute past 3 months? 0 = yes 2 = no | disease in the | 0.0 = less than 3 cups<br>0.5 = 3 to 5 cups<br>1.0 = more than 5 cups | |
| E Neuropsychological problems | | N Mode of feeding | ــــــــــــــــــــــــــــــــــــــ |
| 0 = severe dementia or depression<br>1 = mild dementia<br>2 = no psychological problems | | 0 = unable to eat without assistance<br>1 = self-fed with some difficulty<br>2 = self-fed without any problem | |
| F Body Mass Index (BMI) = weight in kg / (hei<br>0 = BMI less than 19<br>1 = BMI 19 to less than 21<br>2 = BMI 21 to less than 23<br>3 = BMI 23 or greater | ght in m)² | O Self view of nutritional status 0 = views self as being malnourishe 1 = is uncertain of nutritional state 2 = views self as having no nutrition | |
| Screening score (subtotal max. 14 points) | | P In comparison with other people the patient consider his / her heal | |
| 12-14 points: Normal nutritional status 8-11 points: At risk of malnutrition | | 0.0 = not as good<br>0.5 = does not know<br>1.0 = as good | |
| 0-7 points: Malnourished For a more in-depth assessment, continue with q | uestions G-R | 2.0 = better | |
| Assessment | | Q Mid-arm circumference (MAC) in a<br>0.0 = MAC less than 21<br>0.5 = MAC 21 to 22 | cm |
| G Lives independently (not in nursing home of<br>1 = yes 0 = no | | 1.0 = MAC greater than 22 R Calf circumference (CC) in cm | □,□ |
| H Takes more than 3 prescription drugs per d | <br>ay | 0 = CC less than 31<br>1 = CC 31 or greater | П |
| 0 = yes 1 = no | | Assessment (max. 16 points) | |
| I Pressure sores or skin ulcers 0 = yes 1 = no | | Screening score | |
| References 1. Vellas B, Villars H, Abellan G, et al. Overview of the MNA® - Challenges. J Nutr Health Aging. 2006; 10:456-465. 2. Rubenstein LZ, Harker JO, Salva A, Guigoz Y, Vellas B. Scr. Undernutrition in Geriatric Practice: Developing the Short-Fo Nutritional Assessment (MNA-SF). J. Geront. 2001; 56A: M3 3. Guigoz Y. The Mini-Nutritional Assessment (MNA®) Review does it tell us? J Nutr Health Aging. 2006; 10:466-487. | eening for<br>m Mini<br>66-377<br>of the Literature - What | Malnutrition Indicator Score 24 to 30 points 17 to 23.5 points Less than 17 points | Normal nutritional status At risk of malnutrition Malnourished |
| ® Société des Produits Nestlé, S.A., Vevey, Switzerland, Trade | mark Owners | | |



### **CHARLSON INDEX**

| Charlson comorbidity score weights | |
|---|---|
| Charlson Disease category | Original Charlson<br>weights<br>(Charlson,1987) |
| 1. Myocardial Infarction | 1 |
| 2. Congestive heart failure | 1 |
| Peripheral vascular disease | 1 |
| 4. Cerebrovascular disease | 1 |
| 5. Dementia | 1 |
| 6. Chronic pulmonary disease | 1 |
| 7. Rheumatologic disease | 1 |
| 8. Peptic ulcer disease | 1 |
| 9. Mild liver disease | 1 |
| 10. Diabetes | 1 |
| 11. Diabetes with chronic complications | 2 |
| 12. Hemiplegia or paraplegia | 2 |
| 13. Renal disease | 2 |
| 14. Any malignancy, including lymphoma and leukemia | 2 |
| 15. Moderate or severe liver disease | 3 |
| 16. Metastatic solid tumor | 6 |
| 17. AIDS | 6 |
| Maximum Charlson<br>comorbidity score a patient<br>can have | 33 |

Other important medical history:

| • | Hypertension | ( yes / no) |
|---|----------------|-------------|
| • | Dyslipidemia | ( yes / no) |
| • | Osteoarthritis | ( yes / no) |
| • | Mayor surgery | ( yes / no) |
| • | Others: | |



Short-term mortality predictor (< 3 years): score of 0: (12% mortality/year); score 1-2: (26%); score 3-4: (52%); score > 5: (85%).



#### PAIN ASSESMENT ACCORDING TO VAS SCALE:





## COGNITIVE IMPAIRMENT, EMOTIONAL AND RISK OF DELIRIUM ASSESMENT:

### **MINIMENTAL TEST (MMSE):**

| MARCI | Date of Examir | nation | Examiner | | Years of | |
|---|---|---|---|---|---|---|
| | Name | | | Age | | |
| appear in pare<br>Circle 0 if the | ntheses. Administrat | ion should be c<br>, or 1 if the resp | onducted privately<br>oonse is correct. Be | and in the examing gin by asking the fo | minee. Item substitut<br>ee's primary language<br>ollowing two question<br>as about your memo | ns: |
| ORIENTATIO | N TO TIME | , | | RESPONSE | | ORE<br>le one) |
| What is the | year? | | | | 0 | 1 |
| What is the | season? | | | \$0.000 miles | | 1 |
| | month of the year | 2 | | | | 1 |
| | day of the week? | | | | | 1 |
| | date? | | | | | 1 |
| | N TO PLACE* | | | | | |
| Where are we n | now? What is the state (province)? | | | | 0 | 1 |
| | county (or city/town | 1)? | | | | 1 |
| | | | | | 7.0 | 1 |
| | building (name or | and the second s | | | | 1 |
| | floor of the building | 100 | 21- | | 0 | 1 |
| | (room number or ac | | | | | |
| *Alternative place | words that are appropriat | e for the setting an | d increasingly precise r | nay be substituted and | noted. | |
| REGISTRATIC | N* | | | | | |
| Here they are | I am going to say<br>APPLE [pause], PEI<br>times, but score only<br>APPLE | NNY [pause], TA | BLE [pause]. Now | | s back to me. | 1 |
| | PENNY | | | | | 1 |
| ¥ | TABLE | | - | ar ar | 0 | 1 |
| | e words in mind. I a | | | | | |
| ATTENTION | AND CALCULATION | ON [Serial 7s] | * | | | |
| | u to subtract 7 from | | | n each answer unti | I I tell you to stop. | |
| What is 100 tak | | [93] | 3 | | 0 | 1 |
| If needed, say: I | and the same of th | [86] | - | | 0 | 1 |
| If needed, say: I | | [79] | - | | | 1 |
| If needed, say: I | | [72] | | | 0 | 1 |
| If needed, say: I | | [65] | -16 | in State | 0 | 1 |
| A CONTRACTOR OF THE PARTY OF TH | WORLD backward) show | | | | | • |



Substitute and score this item only if the examinee refuses to perform the Serial 7s task.

| Alert/ Drowsy Stuporous C | Comatose/ | | |
|---|---|---|---|
| Assessment of level of consciousness. | (Sum all item scores.) | (30 poir | nts max. |
| | Total Score = | | |
| Score 1 point if the drawing consists of two 5-sided figures th | at rotersect to form a 4-sided figure. | | |
| Please copy this design. [Display the intersecting per | | 0 | 1 |
| DRAWING | | | |
| he sentence is comprehensible and contains a subject and a | verb. Ignore errors in grammar or spening. | | |
| Place the blank piece of paper (unfolded) in front of the exa | | | |
| Please write a sentence. [If examinee does not respon | | 0 | 1 |
| WRITING | | | |
| CLOSE YOUR EYES | | 0 | 1 |
| Please read this and do what it says. [Show examine | ee the words on the stimulus form.] | | |
| READING | | | |
| . TOT ON LOOM (OF TABLE) | | U | |
| PUT ON FLOOR (or TABLE) | | 0 | 1 |
| FOLD IN HALF | | 0 | 1 |
| TAKE IN RIGHT HAND | , | 0 | 1 |
| Listen carefully because I am going to ask you to do<br>Fake this paper in your right hand [pause], fold it in h | | | |
| COMPREHENSION | | | |
| of the page as a stimulus form for the Reading ("CLOSE YO | OUR EYES") and Drawing (intersecting pentagons) if | ems. | |
| the upper half of the page (blank) for the Comprehension, | | | |
| Detach the next page along the lengthwise perforation, and | | | |
| NO IFS, ANDS, OR BUTS. | | 0 | 1 |
| Repeat up to 5 times, but score only the first trial.] | | | |
| Now I am going to ask you to repeat what I say. Read | ly? "NO IFS, ANDS, OR BUTS." Now you say tha | at. | |
| REPETITION | | | |
| Alternative common objects (e.g., eyeglasses, chair, keys) may be | substituted and noted. | | |
| What is this? [Point to a watch.] | 1 2 1 1 1 1 | 0 | 1 |
| What is this? [Point to a pencil or pen.] | 7 | 0 | 1 |
| NAMING* | | 0 | 4 |
| TABLE | | 0 | 1 |
| PENNY | | 0 | 1 |
| APPLE | | 0 | 1 |
| What were those three words I asked you to rememb | er? [Do not offer any hints.] | (circl | e one) |
| RECALL | RESPONSE | | ORE |
| | (D=1) $(L=1)$ $(R=1)$ $(O=1)$ $(W=1)$ | (0 t | 05) |
| out score only the backward spelling. | (D 1) (L 1) (D 1) (O 1) (NL 1) | 10. | - 5) |
| | | _ | |



## **CLOSE YOUR EYES**





### ANEXO 3

## Patient's information obtained from his/her clinical record (Baseline)

| 1. | Patient's ID: | |
|---|---|---|
| 2. | (Register the generic names and total daily dose of drugs that taken during the last month) | t the patient has |
| | Name generic drugs | Total daily<br>dose<br>(milligrams) |



#### 3. **3. Hospitalization**

What was the main cause of hospitalization?

| Diagnosis<br>related<br>Code Group<br>(GRD) | GRD description | Mean stay<br>(days) |
|---|---|---|



## Questionnaire for the subject(baseline)

| 1. | Identification number |
|---|---|
| 2. | Level of studies completed |
| | oCan read and write o Primary o Secondary o University o None |
| 3. | Is the place where you live of your property? |
| | o Yes o No |
| <b>4.</b> | Number of household members where the subject lives: |
| 5. | Carer |
| | a. Do you need a carer to assist you with your daily<br>activities? (for basic hygiene, to help you to move,<br>administration of drugs, performing treatments, etc.Monitoring<br>and supervision tasks are also included) |
| | o Yes o No $\Rightarrow$ Skip to question #6 |
| | <ul> <li>b. In the case of yes, who is your <u>principal carer</u>?</li> <li>o Family member ⇒ Fill in the carer questionnaire and skip to question #6</li> </ul> |
| | o Another non-contracted person (friend) $\Rightarrow$ Fill in the carer questionnaire and skip to question #6 |
| | o Professional carer (contracted or provided by an entity) |
| | c. If you use the services of a <u>professional carer</u> , |
| | How many hours a week? hours a week |
| | Who pays for the service and how much? |
| | o I pay the entire cost of € per hour |
| (Alter | native, if the subject does not know the cost per hour) |



| | o I pay the | entire cost of | € per month |
|---|---|---|---|
| | o The cost | is covered by socia | al security or another entity |
| | | is partially covered<br>€ per hour | d by social security or another entity, I |
| (Alter | native, if the | subject does not k | now the cost per hour) |
| pay _ | o The cost<br>€ per | • | d by social security or another entity, I |
| 6. | Hospitalisa | tion | |
| | Have you | u <u>been admitted t</u> | to hospital in the last 12 months? |
| | o Yes | o No | |

# 7. Health and social services you have required and days of service received by according to economic system during the <u>last month and the last 6 months</u>.

Mark the services you have required, number of days received and form of payment. In case you have required a service and have not received it, note the reason number (see the possible reasons below the table).

| Kinds of services | You<br>have<br>needed<br>to<br>receive | Days service received according to economic system | | | Reason<br>for which<br>they have |
|---|---|---|---|---|---|
| | | Free of charge | Direct<br>paymen<br>t | Mixed<br>(public<br>and<br>private) | not<br>received<br>the<br>service (*) |
| During the <u>last month</u> | | During | | | |
| 1. Telecare | | ——<br>days | days | days | |



| 2. | Domiciliary care /help | days | days | ——<br>days |
|---|---|---|---|---|
| 3. | Day centre | days | days | ——<br>days |
| 4. | Occupational centre or centre for cultural, recreational and leisure activities | days | days | <br>days |
| 5. | Other: | <br>days | days | ——<br>days |
| In | the <u>last 6 months</u> | In the ! | ast 6 mo | <u>nths</u> |
| <b>In</b> 6. | Respite services: Temporary stays | In the I | ast 6 mor | nths<br>days |
| | Respite services: Temporary | | | |

<sup>(\*)</sup> Reasons: 1 – Waiting list. 2 – Not available in the setting. 3 – Cannot pay it. 4 – Does not comply with any of the requirements. 5 – Other reasons.



## QUESTIONNAIRE FOR THE CARER (first contact-baseline)

The subject's principal informal carer (NOT CONTRACTED) fills in the questionnaire.

patient's emotional environment.

The principal informal carer is the person who is in charge of the patient whose autonomy has been limited for health reasons, and the person who spends more time with him/her or who has a greater responsibility to him/her compared with the other members of the

| 1. Identification number: | | | | |
|---|---|---|---|---|
| 2. Carer's | 2. Carer's date of birth (day/month/year): | | | |
| 3. Sex: | | | | |
| o Fei | male | | | |
| o Ma | ale | | | |
| 4. Country | y: | | | |
| 5. Nationa | ality: _ | | | |
| 6. Marita | l status | <b>6:</b> | | |
| o Sin | ngle | o Married or cohabiting | o Divorced | o Separated |
| o Wie | dow | oN/A | | |
| 7. Level | of stud | lies completed: | | |
| o Prim | nary | o Secondary o University | o None | |
| 8. What is | s your ı | elationship with the su | ubject? Are | you his/her |
| o Sib<br>Frien | _ | o Grandchildo Son/daug | hter o Nep | hew/niece o |
| o Ne | ighbour | o Another (please specify | y) | _o N/A |


#### 9. Do you live with the care recipient?

o Yes oNo

#### 10. Since when have you cared for the subject?

O Less than 1 year o between 4 and 6 years

O between 1 and 2 years o More than 6 years

O between 2 and 4 years o NA

#### **HEALTH RELATED PROBLEMS**

- 11. Have you had any health-related problem for caring the subject in the last 12 months?
  - o YES
  - o NO → skip to question #13
- 12. In case of YES, please specify if you suffer any or some of the following problems (multiple choice option):
  - o I am depressed
  - o I am in treatment because of caregiving
  - o I am extremely tired
  - o I have back pain

#### **WORK-RELATED PROBLEM**

#### 13. What is your MAIN working situation?

- o I am employed
- o I am unemployed



| | o Retir | ed or pensione | $ ho r \Rightarrow$ Skip to question #16 |
|---|---|---|---|
| | o Dom | estic tasks ⇒ S | Skip to question #17 |
| | o N/A = | ⇒ Skip to ques | tion #17 |
| | - | - | ork-related problem for caring the subject in |
| τι | | 12 months? | |
| | o Ye | S | o No ⇒ Skip to question #16 |
| 15. | In ca | se of yes, ple | ase specify this |
| | οΙr | equested c | days leave of absence |
| | οΙν | vas working | hours less a day for days |
| | o I a | m working | _ hours less a day |
| | | do not work le | ss hours a day but I have problems fulfilling my |
| | οΙh | ad to leave wo | ork because of illness the person I care |
| | o Ot | her problems: | |
| | etireme<br>ensione | • | e answered in case the carer is retired or a |
| | a. Hav | e you had to | retire early to care for the subject? |
| | o Ye | S | o No $\Rightarrow$ Skip to question #17 |
| | | | lease specify: |
| | οΙr | etired early at | the age of years |



#### **SOCIAL, FAMILY AND LEISURE TIME- RELATED PROBLEMS**

# 17. Have you had any family, social o leisure time-related problem for caring the subject in the last 12 months?

o Yes o No  $\Rightarrow$  Skip to question #19

- **18. In case of YES, please specify this**(multiple choice option):
  - oI had to reduce my leisure time
  - o I have conflicts with my partner or my family
  - o I have no time to see or visit my friends
  - o I have no time to take care of myself or other people
- o I have failed to start a family / I have not been able to have children (or more children)

#### Regarding the role played by you as PRINCIPAL CARER...

| 19. How much time do you invest in a normal DAY for each one of the activities? | | | |
|---|---|---|---|
| Please specify the approximate time you spend <u>daily</u> on each activity | | | |
| On basic hygiene and dressing or changing them | hours | minutes | a day |
| On bathing or showering them | hours | minutes | a day |
| On feeding them | hours | minutes | a day |
| On helping them to move around within the house | hours | minutes | a day |



| On cooking and preparing meals | | hours | | minutes | a day |
|---|---|---|---|---|---|
| Administration of drugs | | hours | | minutes | a day |
| 20. How much time do you invest in a following activities? | norma | al Wi | EEK or | n each oi | ne of the |
| Please specify the approximate time you spend <u>weekly</u> on | each act | ivity | | | |
| On helping them to travel outside the house | | hours | | minutes | a week |
| On helping them to contact health care suppliers | | hours | | minutes | a week |
| On helping them to organise home adaptations | | hours | | minutes | a week |
| On shopping | | hours | | minutes | a week |
| On financial, administrative or legal affairs | | hours | | minutes | a week |
| On social and leisure activities | | hours | | minutes | a week |
| Monitoring and supervision (falls) | | hours | | minutes | a week |

## Regarding the role played by OTHER CARERS (e.g. the rest of the family)

| 21. How much time in a normal DAY dependence of the following activities? Please specify the approximate time these people spend of the spendence of the spend | | - | pend on | each one of |
|---|---|---|---|---|
| On basic hygiene and dressing or changing them | <br>hours | | minutes | a day |
| On bathing or showering them | <br>hours | | minutes | a day |
| On feeding them | <br>hours | | minutes | a day |



| On helping them to move around within the house | | hours | | minutes | a day |
|---|---|---|---|---|---|
| On cooking and preparing meals | | hours | | minutes | a day |
| Administration of drugs | | hours | | minutes | a day |
| 22. How much time do other carers sp following activities? | end ir | n a no | ormal | WEEK ( | on each of the |
| Please specify the approximate time these people spend $\underline{v}$ | <u>veekly</u> on | each a | activity | | |
| On helping them to travel outside the house | | hours | | minutes | a week |
| On helping them to contact health care suppliers | | hours | | minutes | a week |
| On helping them to organise home adaptations | | hours | | minutes | a week |
| On shopping | | hours | | minutes | a week |
| On financial, administrative or legal affairs | | hours | | minutes | a week |
| On social and leisure activities | | hours | | minutes | a week |
| Monitoring and supervision (falls) | | hours | | minutes | a week |



## **QUESTIONNAIRE FOR THE CARER (week 12)**

The subject's principal informal carer (NOT CONTRACTED) fills in the questionnaire

\*If it is the first contact that the care has with the study because the person that she/he looks after did not need a carer before or it is a different carer, the carer must fill the baseline`s questionnaire.

| 1. Identification number |
|---|
| HEALTH RELATED PROBLEMS |
| 2. Have you had any health-related problem for caring the subject in the last 3 months? |
| o YES |
| o NO → skip to question #4 |
| 3. In case of YES, please specify this(multiple choice option):: |
| o I am depressed |
| o I am in treatment because of caregiving |
| o I am extremely tired |
| o I have back pain |
| WORK-RELATED PROBLEM |

4. WHAT IS YOUR MAIN WORKING SITUATION?

o I am employed

78



| | 0 | I am unemployed | |
|---|---|---|---|
| | 0 | Retired or pensioner = | Skip to question #7 |
| | 0 | Domestic tasks $\Rightarrow$ Skip | to question #8 |
| | 0 | $N/A \Rightarrow$ Skip to question | ו #8 |
| 5. | Hav | ve you had any work- | related problem for caring the subject in |
| | the | last 3 months? | |
| | | o Yes | o No $\Rightarrow$ Skip to question #8 |
| 6. | In c | ase of yes, please sp | ecify this |
| | | - , | • |
| | | o I requested days | s leave or absence |
| | | o I was working h | ours less a day for days |
| | | o I am working h | ours less a day |
| | | o I do not work less l<br>working hours | nours a day but I have problems fulfilling my |
| | | o I had to leave work | because of illness the person I care |
| | | o Other problems: | |
| 7. | | irement (only to be a<br>sioner) | nswered in case the carer is retired or a |
| | c. | Have you had to ret | ire early to care for the subject? |
| | | o Yes | o No $\Rightarrow$ Skip to question #8 |
| | d. | In case of yes, pleas | se specify: |
| | | o I retired early at the | e age of years |



#### SOCIAL, FAMILY AND LEISURE TIME- RELATED PROBLEMS

8. Have you had any family, social o leisure time-related problem for caring the subject in the last 3 months?

o Yes

o No  $\Rightarrow$  Skip to question #10

- 9. In case of YES, please specify this(multiple choice option)::
  - oI had to reduce my leisure time
  - o I have conflicts with my partner or my family
  - o I have no time to see or visit my friends
  - o I have no time to take care of myself or other people
- o I have failed to start a family / I have not been able to have children (or more children)

#### Regarding the role played by you as PRINCIPAL CARER...

| 10. How much time do you invest in a normal DAY for each one of the activities? | | | | |
|---|---|---|---|---|
| Please specify the approximate time you spend <u>daily</u> on ea | Please specify the approximate time you spend <u>daily</u> on each activity | | | |
| On basic hygiene and dressing or changing them | | hours | minutes | a day |
| On bathing or showering them | | hours | minutes | a day |
| On feeding them | | hours | minutes | a day |
| On helping them to move around within the house | | hours | minutes | a day |
| On cooking and preparing meals | | hours | minutes | a day |



| Administration of drugs | <br>hours | | minutes | a day |
|---|---|---|---|---|
| 11. How much time do you invest in a following activities? Please specify the approximate time you spend weekly on | | EEK or | ı each o | ne of the |
| On helping them to travel outside the house | <br>hours | | minutes | a week |
| On helping them to contact health care suppliers | <br>hours | | minutes | a week |
| On helping them to organise home adaptations | <br>hours | | minutes | a week |
| On shopping | <br>hours | | minutes | a week |
| On financial, administrative or legal affairs | <br>hours | | minutes | a week |
| On social and leisure activities | <br>hours | | minutes | a week |
| Monitoring and supervision (falls) | <br>hours | | minutes | a week |



#### Regarding the role played by OTHER CARERS (e.g. the rest of the family)

12. How much time in a normal DAY do other carers spend on each one of

| the following activities? | | | | | |
|---|---|---|---|---|---|
| Please specify the approximate time these people spend of | l <u>aily</u> on e | ach act | ivity | | |
| On basic hygiene and dressing or changing them | | hours | | minutes | a day |
| On bathing or showering them | | hours | | minutes | a day |
| On feeding them | | hours | | minutes | a day |
| On helping them to move around within the house | | hours | | minutes | a day |
| On cooking and preparing meals | | hours | | minutes | a day |
| Administration of drugs | | hours | | minutes | a day |
| 13. How much time do other carers sp following activities? Please specify the approximate time these people spend verified to the specifical description of the specifical description. | | | | WEEK oi | n each of the |
| On helping them to travel outside the house | | hours | | minutes | a week |
| On helping them to contact health care suppliers | | hours | | minutes | a week |
| On helping them to organise home adaptations | | hours | | minutes | a week |
| On shopping | | hours | | minutes | a week |
| On financial, administrative or legal affairs | | hours | | minutes | a week |
| On social and leisure activities | | hours | | minutes | a week |



|--|



## **QUESTIONNAIRE FOR THE CARER(week 52)**

The subject's principal informal carer (NOT CONTRACTED) fills in the questionnaire

\*If it is the first contact that the care has with the study because the person that she/he looks after did not need a carer before or it is a different carer, the carer must fill the baseline`s questionnaire.

| 1. Identification number |
|---|
| HEALTH RELATED PROBLEMS |
| 2. Have you had any health-related problem for caring the subject in the last 6 months? |
| o YES |
| o NO $\rightarrow$ skip to question #4 |
| 3. In case of YES, please specify this (multiple choice option):: |
| o I am depressed |
| o I am in treatment because of caregiving |
| o I am extremely tired |
| o I have back pain |
| o I have no problem of health because of caregiving |

#### **WORK-RELATED PROBLEM**



| 4 | MAZILAT TO | VALID | | WODISTNIC | CTTLLATIONS |
|----|------------|-------|------|-----------|-------------|
| 4. | WHAI 15 | YOUK | MAIN | WORKING | SITUATION? |

| o I am employed o I am unemployed o Retired or pensioner ⇒ Skip to question #7 o Domestic tasks ⇒ Skip to question #8 o N/A ⇒ Skip to question #8 5. Have you had any work-related problem for caring the subject if the last 6 months? o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling materials working hours o I had to leave work because of illness the person I care o Other problems: | | |
|---|---|---|
| o Retired or pensioner ⇒ Skip to question #7 o Domestic tasks ⇒ Skip to question #8 o N/A ⇒ Skip to question #8 5. Have you had any work-related problem for caring the subject if the last 6 months? o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | o I am employed |
| o Domestic tasks ⇒ Skip to question #8 o N/A ⇒ Skip to question #8 5. Have you had any work-related problem for caring the subject if the last 6 months? o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | o I am unemployed |
| o N/A ⇒ Skip to question #8 5. Have you had any work-related problem for caring the subject if the last 6 months? o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | o Retired or pensioner $\Rightarrow$ Skip to question #7 |
| <ul> <li>5. Have you had any work-related problem for caring the subject if the last 6 months?</li> <li>o Yes</li> <li>o No ⇒ Skip to question #8</li> <li>6. In case of yes, please specify this</li> <li>o I requested days leave of absence</li> <li>o I was working hours less a day for days</li> <li>o I am working hours less a day</li> <li>o I do not work less hours a day but I have problems fulfilling morking hours</li> <li>o I had to leave work because of illness the person I care</li> </ul> | | o Domestic tasks $\Rightarrow$ Skip to question #8 |
| the last 6 months? o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | o N/A $\Rightarrow$ Skip to question #8 |
| the last 6 months? o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | |
| o Yes o No ⇒ Skip to question #8 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | 5. | |
| 6. In case of yes, please specify this o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | the last 6 months? |
| o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling morking hours o I had to leave work because of illness the person I care | | o Yes o No $\Rightarrow$ Skip to question #8 |
| o I requested days leave of absence o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling morking hours o I had to leave work because of illness the person I care | | |
| o I was working hours less a day for days o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | 6. | In case of yes, please specify this |
| o I am working hours less a day o I do not work less hours a day but I have problems fulfilling m working hours o I had to leave work because of illness the person I care | | o I requested days leave of absence |
| o I do not work less hours a day but I have problems fulfilling m<br>working hours<br>o I had to leave work because of illness the person I care | | o I was working hours less a day for days |
| working hours o I had to leave work because of illness the person I care | | o I am working hours less a day |
| | | o I do not work less hours a day but I have problems fulfilling mover working hours |
| o Other problems: | | o I had to leave work because of illness the person I care |
| | | o Other problems: |

## 7. Retirement (only to be answered in case the carer is retired or a pensioner)

e. Have you had to retire early to care for the subject?

o Yes o No  $\Rightarrow$  Skip to question #8



| f. | In | case | of yes | , please | specify: |
|----|----|------|--------|----------|----------|
|----|----|------|--------|----------|----------|

o I retired early at the age of\_\_\_\_ years

#### SOCIAL, FAMILY AND LEISURE TIME- RELATED PROBLEMS

8. Have you had any family, social o leisure time-related problem for caring the subject in the last 6 months?

o Yes o No  $\Rightarrow$  Skip to question #10

- **9.** In case of YES, please specify this (multiple choice option):
  - o I had to reduce my leisure time
  - o I have conflicts with my partner or my family
  - o I have no time to see or visit my friends
  - o I have no time to take care of myself or other people
- o I have failed to start a family / I have not been able to have children (or more children)

#### Regarding the role played by you as PRINCIPAL CARER...

| 10. How much time do you invest in a normal DAY for each one of the activities? | | | |
|---|---|---|---|
| Please specify the approximate time you spend <u>daily</u> on each activity | | | |
| On basic hygiene and dressing or changing them | hours | minutes | a day |
| On bathing or showering them | hours | minutes | a day |



| On feeding them | | hours | | minutes | a day |
|---|---|---|---|---|---|
| On helping them to move around within the house | | hours | | minutes | a day |
| On cooking and preparing meals | | hours | | minutes | a day |
| Administration of drugs | | hours | | minutes | a day |
| 11. How much time do you invest in a normal WEEK on each one of the following activities? | | | | | |
| following activities? | | | EEK oı | n each o | ne of the |
| | | | EEK oı | n each o | ne of the |
| following activities? | | | EEK oi | minutes | ne of the |
| following activities? Please specify the approximate time you spend weekly on | | tivity | EEK oi | | |
| following activities? Please specify the approximate time you spend weekly on On helping them to travel outside the house | each act | hours | | minutes | a week |

hours

hours

hours

minutes

minutes

minutes

a week

a week

a week

On financial, administrative or legal affairs

On social and leisure activities

Monitoring and supervision (falls)



#### Regarding the role played by OTHER CARERS (e.g. the rest of the family)

12. How much time in a normal DAY do other carers spend on each one of

| the following activities? | | | | | |
|---|---|---|---|---|---|
| Please specify the approximate time these people spend <u>daily</u> on each activity | | | | | |
| On basic hygiene and dressing or changing them | | hours | | minutes | a day |
| On bathing or showering them | | hours | | minutes | a day |
| On feeding them | | hours | | minutes | a day |
| On helping them to move around within the house | | hours | | minutes | a day |
| On cooking and preparing meals | | hours | | minutes | a day |
| Administration of drugs | | hours | | minutes | a day |
| 13. How much time do other carers spend in a normal WEEK on each of the following activities? Please specify the approximate time these people spend weekly on each activity | | | | | |
| riease specify the approximate time these people spend v | VEEKIY OII | Cacire | ictivity | | |
| On helping them to travel outside the house | | hours | | minutes | a week |
| On helping them to contact health care suppliers | | hours | | minutes | a week |
| On helping them to organise home adaptations | | hours | | minutes | a week |
| On shopping | | hours | | minutes | a week |
| On financial, administrative or legal affairs | | hours | | minutes | a week |
| On social and leisure activities | | hours | | minutes | a week |



| Г |
|---|



#### 12. REFERENCES

- 1. Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, et al. Frailty in older adults: evidence for a phenotype. The journals of gerontology Series A, Biological sciences and medical sciences. 2001;56(3):M146-56.
- 2. Ferrucci L, Cavazzini C, Corsi A, Bartali B, Russo CR, Lauretani F, et al. Biomarkers of frailty in older persons. Journal of endocrinological investigation. 2002;25(10 Suppl):10-5.
- 3. Fried LP, Guralnik JM. Disability in older adults: evidence regarding significance, etiology, and risk. Journal of the American Geriatrics Society. 1997;45(1):92-100.
- 4. Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Archives of internal medicine. 2006;166(4):418-23.
- 5. Xue QL. The frailty syndrome: definition and natural history. Clinics in geriatric medicine. 2011;27(1):1-15.
- 6. Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, et al. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. Jama. 2014;311(23):2387-96.
- 7. Gill TM, Gahbauer EA, Han L, Allore HG. Trajectories of disability in the last year of life. The New England journal of medicine. 2010;362(13):1173-80.
- 8. Sourial N, Bergman H, Karunananthan S, Wolfson C, Payette H, Gutierrez-Robledo LM, et al. Implementing frailty into clinical practice: a cautionary tale. The journals of gerontology Series A, Biological sciences and medical sciences. 2013;68(12):1505-11.
- 9. Bandeen-Roche K, Xue QL, Ferrucci L, Walston J, Guralnik JM, Chaves P, et al. Phenotype of frailty: characterization in the women's health and aging studies. The journals of gerontology Series A, Biological sciences and medical sciences. 2006;61(3):262-6.
- 10. Garcia-Garcia FJ, Gutierrez Avila G, Alfaro-Acha A, Amor Andres MS, De Los Angeles De La Torre Lanza M, Escribano Aparicio MV, et al. The prevalence of frailty syndrome in an older population from Spain. The Toledo Study for Healthy Aging. The journal of nutrition, health & aging. 2011;15(10):852-6.
- 11. Campbell AJ, Buchner DM. Unstable disability and the fluctuations of frailty. Age and ageing. 1997;26(4):315-8.
- 12. Walston J, Fried LP. Frailty and the older man. The Medical clinics of North America. 1999;83(5):1173-94.
- 13. Rockwood K, Hogan DB, MacKnight C. Conceptualisation and measurement of frailty in elderly people. Drugs & aging. 2000;17(4):295-302.
- 14. Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013;381(9868):752-62.
- 15. Strandberg TE, Pitkala KH. Frailty in elderly people. Lancet. 2007;369(9570):1328-9.
- 16. Rodriguez-Artalejo F, Rodriguez-Manas L. The frailty syndrome in the public health agenda. Journal of epidemiology and community health. 2014;68(8):703-4.
- 17. Barnett K, Mercer SW, Norbury M, Watt G, Wyke S, Guthrie B. Epidemiology of multimorbidity and implications for health care, research, and medical education: a cross-sectional study. Lancet. 2012;380(9836):37-43.
- 18. Temple RM, Kirthi V, Patterson LJ. Is it time for a new kind of hospital physician? Bmj. 2012;344:e2240.
- 19. Stuck AE, Iliffe S. Comprehensive geriatric assessment for older adults. Bmj. 2011;343:d6799.



- 20. Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, et al. Frailty assessment in the cardiovascular care of older adults. Journal of the American College of Cardiology. 2014;63(8):747-62.
- 21. Balducci L, Colloca G, Cesari M, Gambassi G. Assessment and treatment of elderly patients with cancer. Surgical oncology. 2010;19(3):117-23.
- 22. Ellis G, Whitehead MA, Robinson D, O'Neill D, Langhorne P. Comprehensive geriatric assessment for older adults admitted to hospital: meta-analysis of randomised controlled trials. Bmj. 2011;343:d6553.
- 23. Partridge JS, Harari D, Dhesi JK. Frailty in the older surgical patient: a review. Age and ageing. 2012;41(2):142-7.
- 24. Philipps V, Amieva H, Andrieu S, Dufouil C, Berr C, Dartigues JF, et al. Normalized Mini-Mental State Examination for assessing cognitive change in population-based brain aging studies. Neuroepidemiology. 2014;43(1):15-25.
- 25. Morley JE. Developing novel therapeutic approaches to frailty. Current pharmaceutical design. 2009;15(29):3384-95.
- 26. Mahoney FI, Barthel DW. Functional Evaluation: The Barthel Index. Maryland state medical journal. 1965;14:61-5.
- 27. Yesavage JA. Geriatric Depression Scale. Psychopharmacology bulletin. 1988;24(4):709-11.
- 28. Sinclair AJ, Armes DG, Randhawa G, Bayer AJ. Caring for older adults with diabetes mellitus: characteristics of carers and their prime roles and responsibilities. Diabetic medicine : a journal of the British Diabetic Association. 2010;27(9):1055-9.
- 29. Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Annals of internal medicine. 1990;113(12):941-8.
- 30. Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, et al. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. Journal of gerontology. 1994;49(2):M85-94.
- 31. Schuit AJ, Schouten EG, Westerterp KR, Saris WH. Validity of the Physical Activity Scale for the Elderly (PASE): according to energy expenditure assessed by the doubly labeled water method. Journal of clinical epidemiology. 1997;50(5):541-6.
- 32. Vellas B, Villars H, Abellan G, Soto ME, Rolland Y, Guigoz Y, et al. Overview of the MNA-lts history and challenges. The journal of nutrition, health & aging. 2006;10(6):456-63; discussion 63-5.
- 33. Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. Journal of chronic diseases. 1987;40(5):373-83.
- 34. Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011;152(10):2399-404.
- 35. Bermejo F, Morales JM, Valerga C, del Ser T, Artolazabal J, Gabriel R. [A comparison between 2 abbreviated Spanish versions of mental status assessment in the diagnosis of dementia. Study data on elderly community residents]. Medicina clinica. 1999;112(9):330-4.